CLINICAL TRIAL: NCT06693011
Title: Contour Neurovascular System™ ContiNued Access Investigational Device EXempTion (IDE) Trial
Brief Title: Contour Neurovascular System™ ContiNued Access Investigational Device EXempTion (IDE) Trial (NEXT Trial)
Acronym: NEXT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cerus Endovascular, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DNX140-01
Record Dates: First submitted 2024-11-08; First posted 2024-11-18 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-07

CONDITIONS: Cerebral Aneurysms
Keywords: aneurysm; wide-neck; bifurcated; saccular
MeSH Terms: conditions — Intracranial Aneurysm; Aneurysm

STUDY DESIGN:
Intervention Model Description: This study is a prospective, multicenter, single-arm study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Treatment Attempt with the Contour Neurovascular System (Experimental): Subjects for which the index procedure (implant of the Contour Neurovascular System) was attempted.
  Interventions: Device: Contour Neurovascular System Treatment Attempt

INTERVENTIONS:
Device: Contour Neurovascular System Treatment Attempt — The subject is brought into the procedure room, an angiogram on the day of the procedure indicates that the subject is anatomically eligible for the trial and any part of the investigational device comes in contact with the patient

SUMMARY:
The goal of this clinical trial is to collect additional data to demonstrate if the Contour Neurovascular System (CNS) is a safe and effective treatment of wide-necked, saccular, intracranial aneurysms.

Participants will:

Undergo treatment with the Contour Neurovascular System Complete follow-up visits at 1month, 12months, and 24 months, following their procedure Report any adverse events to their study team

ELIGIBILITY:
Inclusion Criteria:

1. Patient is 18-75 years of age at the time of screening.
2. Patient has a single ruptured or unruptured IA requiring treatment. If the patient has an additional IA requiring treatment, the additional IA must not require treatment within 60 days after the index procedure.
3. The target IA must have the following characteristics:

   * Saccular morphology
   * Located at a bifurcation in the anterior or posterior circulation
   * Aneurysm neck diameter between 2 and 10 mm and aneurysm equatorial diameter between 2 and 10.5 mm
   * Wide-necked, defined as neck size ≥ 4 mm or a dome/neck ratio < 2
4. Patient may be treated with Contour without the use of additional implanted devices.
5. Patient is able to comply with all aspects of the screening, evaluation, treatment, and the post-procedure follow-up schedule.
6. Patient or legally authorized representative has signed and dated an institutional review board (IRB)/Ethics Committee (EC)-approved written informed consent prior to initiation of any study procedures.

   FOR PATIENTS WITH UNRUPTURED ANEURYSM
7. Patient meets the criteria outlined in the "Guidelines for the Management of Patients With Unruptured Intracranial Aneurysms" as published by the AHA/ASA^6

   FOR PATIENTS WITH RUPTURED ANEURYSM
8. Patient meets the criteria outlined in the "Guidelines for the Management of Aneurysmal Subarachnoid Hemorrhage: A Guideline for Healthcare Professionals from the American Heart Association/American Stroke Association" as published by the AHA/ASA.^6
9. Patient must be neurologically stable with Hunt & Hess Score of I, II or III.

(^6: 6 https://www.ahajournals.org/doi/full/10.1161/STR.0000000000000070)

Exclusion Criteria:

1. Anatomy or physiology considered unsuitable for endovascular treatment with the Contour device by the implanting physician and/or the Patient Selection Committee
2. Target IA contains other devices/implants (e.g., coils) that could interfere with the correct placement of the Contour device
3. Subject has a known, untreatable hypersensitivity to contrast dye, iodine, or any component of the treatment device.
4. Contraindication to anticoagulants or anti-platelet medications
5. Stenosis of the target IA's parent vessel is >50%
6. Anticoagulation medications (e.g., warfarin) that cannot be discontinued
7. Acute / chronic renal failure (unless on dialysis) or creatinine > 2.00 mg/dl or > 182 μmol/L
8. Vascular disease or other vascular anomaly that precluded the necessary access to the aneurysm for use of the study device.
9. Clinical, angiographic or computed tomography (CT) evidence of vasospasm, vasculitis, an intracranial tumor (except small meningioma) or any other intracranial vascular malformations on presentation.
10. Conditions placing them at high risk for ischemic stroke or had exhibited ischemic symptoms such as transient ischemic attacks, minor strokes, or stroke-in-evolution within the prior 60-days.
11. Any circulatory, neurovascular, cardiovascular, or neurologic conditions that can result in unstable neurological symptoms (e.g., multiple sclerosis, established seizure disorder).
12. Modified Rankin Scale (mRS) score ≥ 2 prior to presentation or rupture (as applicable).
13. Subarachnoid hemorrhage (SAH) from a non-index aneurysm or any other intracranial hemorrhage within 90 days.
14. Physical, neurologic or psychiatric conditions which precluded his/her ability to comply with all aspects of the screening, evaluation, treatment, and the post-procedure follow-up schedule.
15. Pregnant, breastfeeding or planning pregnancy in the next 2 years
16. Subject is enrolled in another device or drug study in which participation could confound study results.
17. Life expectancy of less than 2 years due to an illness or condition other than the index intracranial aneurysm.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-06-10 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of death or stroke within 30 days of treatment or ipsilateral stroke or neurological death between 30 days and 1 year. | From enrollment to 1 year
  Death or stroke within 30 days of treatment or ipsilateral stroke or neurological death between 30 days and 1 year.
  Stroke is defined per the World Health Organization as: rapidly developing clinical signs of focal or global disturbance of cerebral function lasting more than 24 hours with no apparent cause other than of vascular origin, including ischemic stroke and/or hemorrhagic stroke.
Proportion of complete occlusion of the aneurysm with Contour, without retreatment, recurrent subarachnoid hemorrhage, or significant parent artery stenosis at one (1) year after treatment. | From enrollment to 1 year
  Complete occlusion of the aneurysm with Contour as defined by complete aneurysm occlusion (Raymond Roy Scale of 1) without retreatment, recurrent subarachnoid hemorrhage, or significant parent artery stenosis (> 50% stenosis) at one (1) year after treatment as assessed by the angiographic core laboratory.
  The Raymond-Roy Scale grades aneurysms on a scale of one (1) to three (3) with a lower score correlating with a more favorable outcome. The Raymond-Roy Scale will be graded in accordance with the following definitions: Class 1 (Complete obliteration of the aneurysm), Class 2 (Persistence of any portion of the original defect of the arterial wall as seen on any single projection but without opacification of the aneurysmal sac), or Class 3 (Any opacification of the aneurysmal sac).

SECONDARY OUTCOMES:
Incidence of Serious Adverse Events (SAE) associated with the procedure or device | From enrollment to 2 years
  Serious Adverse Events (SAE) associated with the procedure or device, both individually and in aggregate
Proportions of aneurysm occlusion ratings | From enrollment to 2 years
  ·Detailed assessment of aneurysm occlusion from post procedure to one (1) year (and also at two (2) years for any aneurysm not completely occluded at 1 year) provided by the core lab review of the angiogram, including the following:
  * Complete occlusion (Raymond Roy Scale of 1)
  * Adequate Occlusion (Raymond Roy Scale of 1 or 2)
  * Raymond Roy scale
  The Raymond-Roy Scale grades aneurysms on a scale of one (1) to three (3) with a lower score correlating with a more favorable outcome. The Raymond-Roy Scale will be graded in accordance with the following definitions: Class 1 (Complete obliteration of the aneurysm), Class 2 (Persistence of any portion of the original defect of the arterial wall as seen on any single projection but without opacification of the aneurysmal sac), or Class 3 (Any opacification of the aneurysmal sac).
Incidence of stroke resulting in a disabling deficit | From enrollment to 2 years
  Assessment of incidence of stroke resulting in a disabling deficit, defined operationally as a deficit that, if unchanged, would prevent the patient from performing basic activities of daily living (i.e., bathing, ambulating, toileting, hygiene, and eating) or returning to work (mRS ≥ 3).
Incidence of serious neurological events | From enrollment to 2 years
  All serious neurological adverse events
Proportions of device movement ratings | From enrollment to 2 years
  ·Detailed assessment of aneurysm occlusion from post procedure to one (1) year (and also at two (2) years for any aneurysm not completely occluded at 1 year) provided by the core lab review of the angiogram, including the following:
  o Device position (remains in place, migration into the parent artery or movement towards the aneurysm dome)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University at Buffalo Neurosurgery, Buffalo, New York
  - Stony Brook University, Stony Brook, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Swedish Neuroscience Institute, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No